CLINICAL TRIAL: NCT05415748
Title: PlacEbo-controlled, Randomized, Patient-Selected Outcomes N-of-1 triALs (PERSONAL-pilot): Alpha-blockers for Lower Urinary Tract Symptoms
Brief Title: Deprescribing Tamsulosin in Older Men
Acronym: PERSONAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-28557; K12DK111028 (NIH)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin 0.4 mg or 0.8 mg, Then Placebo (Experimental): Participants first received Tamsulosin 0.4 mg or 0.8 mg taken daily in 2 week treatment periods, 4 treatment periods in 12 weeks. After a washout period of 1 week, the participants then received Placebo tablet taken daily in 2 week treatment periods, 4 treatment periods in 12 weeks.
  Interventions: Drug: Tamsulosin; Drug: Placebo
- Placebo, Then Tamsulosin 0.4 mg or 0.8 mg (Experimental): Participants first received Placebo tablet taken daily in 2 week treatment periods, 4 treatment periods in 12 weeks. After a washout period of 1 week, the participants then received Tamsulosin 0.4 mg or 0.8 mg taken daily in 2 week treatment periods, 4 treatment periods in 12 weeks.
  Interventions: Drug: Tamsulosin; Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin and matching placebo to be taken in a randomized order for 12 weeks
  Other Names: Flomax
Drug: Placebo — Tamsulosin and matching placebo to be taken in a randomized order for 12 weeks

SUMMARY:
This is a pilot 12-week randomized, placebo-controlled N-of-1 deprescribing trial among older men receiving chronic tamsulosin therapy for lower urinary tract symptoms attributed to benign prostatic hyperplasia.

DETAILED DESCRIPTION:
The investigators will instruct participants to monitor and record their daily urinary symptoms and medication side effects through Redcap surveys, accessible via smartphone. Medication adherence, global urinary satisfaction questions, and health-related quality of life will be assessed as baseline and at the end of the study.

Monitoring frequency: Participants will monitor their symptoms every day using the PERSONAL-pilot study Redcap surveys. If the investigators notice a subject has been unresponsive to daily symptom monitoring, the investigators will reach out to the subject and offer any help we can provide. The investigators first attempt will be in the form of an email, sent to the email address provided to send patients the surveys. If the investigators do not receive a response, the investigators will follow up with a phone call to offer any help or guidance. Email template and telephone script provided in other study documents of the application.

N-of-1 Trial Procedures:

Participants will start with a 1-week open label period where participants will use the PERSONAL Redcap surveys to track daily symptoms and side effects while not taking their tamsulosin or any study pills. Based on the pharmacokinetics and expected timeframe of symptomatic relief from tamsulosin (half-life=14 to 15 hours; steady state by the 5th day of daily dosing), all N-of-1 trials will have a duration of 11 weeks during which participants will complete 2 cycles consisting of a pair of 2-week treatment periods (taking tamsulosin or placebo) separated by 1 week of wash-out on placebo. The order of treatment periods within a cycle will be random (e.g. ABAB, BABA, ABBA, or BAAB) according to pre-filled bubble packs given to participants during their orientation visit.

Participants will receive a placebo during wash-out periods between treatment periods and cycles, but the participants will be unaware of the order or duration of treatment periods or cycles to prevent self-correlating symptoms to specific treatments.

The PERSONAL Redcap will present participants with a daily questionnaire, accessible via smartphone, to track their lower urinary tract symptoms and medication side effects. All participants will also be presented a global urinary symptom bother question. At the end of each week, participants will receive additional medication adherence and treatment satisfaction questionnaires administered via the PERSONAL app as well as motivational messages summarizing their progress in the trial.

Participants will view a graphical representation of their responses summarized in chronological order for the prior day, week, or month. To maximize adherence to daily questionnaires, participants will be contacted via email or phone if they have completed fewer than 4 daily questionnaires in any week during their N-of-1 trial. At the end of the study, the participants will complete an end of-study questionnaire and a 10-30 min. interview with staff member with formal qualitative research training. Then, PERSONAL staff will review N-of-1 trial results with the participant.

ELIGIBILITY:
Inclusion Criteria:

* Urology patient at UCSF
* Must own Android or iPhone smartphone, tablet, or computer
* Taking tamsulosin for urinary-related symptoms
* Able to speak and read English
* Male 55-80 years old of age at telephone screening.
* Written informed consent (and assent when applicable) obtained from subject or subject' s legal representative and ability for subject to comply with the requirements of the study.
* Willing to receive electronic PERSONAL daily intake surveys for 3 months
* Willing to self-report urinary symptom or medication side effect data at specified frequency.
* Have home WiFi access.
* Patients with h/o prostate cancer may be enrolled but is not required
* Patients with h/o kidney stones may be enrolled but is not required

Exclusion Criteria:

* Taking tamsulosin for <12 months.
* International Prostate Symptom Score <5 or >25
* Current participation in any other mobile app-based clinical study.
* Planning to relocate from area within the study duration.
* Impaired vision that could limit the use of the mobile apps (participant-reported)

Ages: 55 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjmain N Breyer, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is their original dosage of either 0.4 or 0.8 mg of tamsulosin and we are showing in the results on the drug or off the drug periods.
Groups:
- Placebo Then Tamsulosin, Placebo Then Tamsulosin: Tamsulosin and matching placebo to be taken in a randomized quarter for 12 weeks after a one-week placebo run-in. After the one week placebo run-in, participants first received placebo taken daily for a 2 week treatment period, followed by a one week placebo washout, followed by tamsulosin 0.4 mg or 0.8 mg taken daily for a two week treatment period, followed by a one week placebo washout, participants then received placebo taken daily for a 2 week treatment period, followed by a one week placebo washout, followed by tamsulosin 0.4 mg or 0.8 mg taken daily for a two week treatment period.
- Placebo Then Tamsulosin, Tamsulosin Then Placebo: Tamsulosin and matching placebo to be taken in a randomized quarter for 12 weeks after a one-week placebo run-in. After the one week placebo run-in, participants first received placebo taken daily for a 2 week treatment period, followed by a one week placebo washout, followed by tamsulosin 0.4 mg or 0.8 mg taken daily for a two week treatment period, followed by a one week placebo washout, participants then received tamsulosin 0.4 mg or 0.8 mg taken daily for a 2 week treatment period, followed by a one week placebo washout, followed by placebo taken daily for a two week treatment period.
- Tamsulosin Then Placebo, Tamsulosin Then Placebo: Tamsulosin and matching placebo to be taken in a randomized quarter for 12 weeks after a one-week placebo run-in. After the one week placebo run-in, participants first received tamsulosin 0.4 mg or 0.8 mg taken daily for a 2 week treatment period, followed by a one week placebo washout, followed by placebo taken daily for a two week treatment period, followed by a one week placebo washout, participants then received tamsulosin 0.4 mg or 0.8 mg taken daily for a 2 week treatment period, followed by a one week placebo washout, followed by placebo taken daily for a two week treatment period
- Tamsulosin Then Placebo, Placebo Then Tamsulosin: Tamsulosin and matching placebo to be taken in a randomized quarter for 12 weeks after a one-week placebo run-in. After the one week placebo run-in, participants first received tamsulosin 0.4 mg or 0.8 mg taken daily for a 2 week treatment period, followed by a one week placebo washout, followed by placebo taken daily for a two week treatment period, followed by a one week placebo washout, participants then received placebo taken daily for a 2 week treatment period, followed by a one week placebo washout, followed by tamsulosin 0.4 mg or 0.8 mg taken daily for a two week treatment period.
Period: Wash-out #1 (1 Week)
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Started | 7 | 8 | 8 | 8
Completed | 6 | 7 | 6 | 8
Not Completed | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0
Period: Intervention #1 (2 Weeks)
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Started | 6 | 7 | 6 | 8
Completed | 6 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out #2 (1 Week)
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Started | 6 | 7 | 6 | 8
Completed | 6 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Intervention #2 (2 Weeks)
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Started | 6 | 7 | 6 | 8
Completed | 5 | 7 | 6 | 8
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Wash-out #3 (1 Week)
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Started | 5 | 7 | 6 | 8
Completed | 5 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Intervention #3 (2 Weeks)
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Started | 5 | 7 | 6 | 8
Completed | 5 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out #4 (1 Week)
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Started | 5 | 7 | 6 | 8
Completed | 5 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Intervention #4 (2 Weeks)
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Started | 5 | 7 | 6 | 8
Completed | 5 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is their original dosage of either 0.4 or 0.8 mg of tamsulosin and we are showing in the results on the drug or off the drug periods.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin | Total
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 31
Age, Customized [Count of Participants; unit: Participants]
  less than 55 | 0 | 0 | 0 | 0 | 0
  over 55, less than 81 | 7 | 8 | 8 | 8 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 8 | 8 | 8 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 5 | 7 | 8 | 7 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Adapted International Prostate Symptom Score (IPSS)
Description: Lower urinary tract symptoms will be measured using the adapted IPSS (recall period changed from 1 month to 24 hours). The score ranges from 0-35, with higher scores indicating more severe symptoms.
Time Frame: Every day for 12 weeks. Daily adapted IPSS scores will be averaged over the treatment period.
Population: A direct comparison between the 0.4 mg and 0.8 mg dose groups was not pre-specified in the study design and was therefore not conducted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Number analyzed (Participants) | 5 | 7 | 6 | 8
score on a scale
  Tamsulosin | 13.5 (9.5) | 12.1 (8.0) | 14.1 (7.5) | 9.2 (6.0)
  Placebo | 18.7 (7.5) | 14.3 (7.9) | 17.6 (6.4) | 10.9 (7.2)

2. Secondary Outcome: Medication Side Effect Scale
Description: It's a self-reported instrument assessing the presence and severity of common tamsulosin side effects over the past 24 hour period. Possible scores range from 0 (not at all bothered) to 3 (extremely bothered). The total score ranges from 0-36.
Time Frame: Daily for 12 weeks. Daily adapted IPSS scores will be averaged over the treatment period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Then Tamsulosin, Placebo Then Tamsulosin | Placebo Then Tamsulosin, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Tamsulosin Then Placebo | Tamsulosin Then Placebo, Placebo Then Tamsulosin
Number analyzed (Participants) | 5 | 7 | 6 | 8
score on a scale
  Tamsulosin | 0.94 (1.24) | 2.59 (1.94) | 1.43 (2.49) | 1.15 (1.47)
  Placebo | 1.27 (1.41) | 2.58 (1.90) | 1.11 (1.62) | 1.20 (1.48)

3. Other Pre Specified Outcome: Urinary Bother Scale
Description: It's a self-reported instrument assessing how the participants would feel if they were to spend the rest of their life with their urinary condition as it is now for the past 24 hour period. Possible scores range from 0 (delighted) to 6 (terrible).
Time Frame: Baseline and 12-week follow-up
Reporting Status: Not Posted

4. Other Pre Specified Outcome: PROMIS 29 v2.0
Description: The PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain.
Time Frame: Baseline and 12-week follow-up
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Voils Medication Adherence Questionnaire
Description: Participants were asked several questions regarding the extent of medication nonadherence and the reasons for medication nonadherence.
  For the extent of medication nonadherence, 3 questions were asked. Possible scores range from 0 (strongly disagree) to 4 (strongly agree, worse outcome) per question.
  For the reasons of medication nonadherence, 19 questions were asked. Possible scores range from 0 (not at all) to 4 (very much, worse outcome) per question.
Time Frame: Baseline and 12-week follow-up
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Post-Study System Usability Questionnaire
Description: Participants were asked their perceived satisfaction with the usability of the PERSONAL app. 8 questions were asked. Possible scores range from 0 (strongly disagree) to 4 (strongly agree, better outcome) per question.
Time Frame: 12-week follow-up
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Revised Patients' Attitudes Towards Deprescribing (rPATD) Questionnaire
Description: Participants were asked several questions regarding their beliefs and attitudes towards deprescribing.
Time Frame: Baseline and 12-week follow-up
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Perceived Change in Urinary Status Questionnaire
Description: Participants were asked several questions if they felt that their urinary symptoms were unchanged, improved, or worsened
Time Frame: Baseline and 12-week follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Placebo/Tamsulosin: Tamsulosin and matching placebo to be taken in a randomized order for 12 weeks. Participants first received Tamsulosin 0.4 mg or 0.8 mg taken daily in 2 week treatment periods, 4 treatment periods in 12 weeks. After a washout period of 1 week, the participants then received Placebo tablet taken daily in 2 week treatment periods, 4 treatment periods in 12 weeks.
Arm/Group | Placebo/Tamsulosin
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT05415748/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT05415748/ICF_001.pdf